CLINICAL TRIAL: NCT07345572
Title: Investigating the Impact of Early Time-Restricted Eating on Health Outcomes and Quality of Life in Adults With and Without Asthma
Brief Title: Investigating the Impact of Early Time-Restricted Eating on Health Outcomes and Quality of Life in Adults With Mild Controlled Asthma Compared to Healthy Adults
Acronym: eTRE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: De Montfort University (Other)
Collaborators: King Saud Bin Abdulaziz University for Health Sciences (Other)
Responsible Party: Principal Investigator, Nouf Alotaibi, Principal Investigator, De Montfort University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LSREF2568554
Record Dates: First submitted 2025-12-03; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Asthma Management; Time Restricted Eating
Keywords: Asthma; time restricted eating; inflammatory markers; oxidative stress markers; pulmonary function parameters; quality of life; adherence
MeSH Terms: conditions — Intermittent Fasting; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Habitual Diet (HD) and early Time Restricted Eating (eTRE) (Active Comparator): The participants will be asked to follow their habitual diet for one week. After two weeks washout period, the participants will be assigned to eTRE and asked to eat from 8 am to 4 pm without restriction on the quantity or amount of food and fast for the rest of the time except for drinking water for one week.
  Interventions: Other: Habitual Diet (HD) and Early Time-Restricted Eating (eTRE)
- early Time Restricted Eating (eTRE) and Habitual Diet (HD) (Active Comparator): The participants who are assigned to eTRE will be asked to eat from 8 am to 4 pm without restriction on the quantity or amount of food and fast for the rest of the time except for drinking water for one week. After two weeks washout period, participants will be asked to follow their habitual diet for one week.
  Interventions: Other: Early Time-Restricted Eating (eTRE) and Habitual Diet (HD)

INTERVENTIONS:
Other: Early Time-Restricted Eating (eTRE) and Habitual Diet (HD) — The participants who are assigned to eTRE will be asked to eat from 8 am to 4 pm without restriction on the quantity or amount of food and fast for the rest of the time except for drinking water for one week. After two weeks washout period, participants will be asked to follow their habitual diet for one week.
  Other Names: eTRE
  Arms: early Time Restricted Eating (eTRE) and Habitual Diet (HD)
Other: Habitual Diet (HD) and Early Time-Restricted Eating (eTRE) — The participants will be asked to follow their habitual diet for one week. After two weeks washout period, the participants will be assigned to eTRE and asked to eat from 8 am to 4 pm without restriction on the quantity or amount of food and fast for the rest of the time except for drinking water for one week.
  Arms: Habitual Diet (HD) and early Time Restricted Eating (eTRE)

SUMMARY:
This study aims to explore how early time-restricted eating (eTRE) - where all daily meals are eaten within a specific time window - affects health and quality of life in adults. The researchers will compare results between adults with mild, well-controlled asthma and adults without asthma (the control group). Participants can continue to eat their normal food; only the timing of meals will change.

DETAILED DESCRIPTION:
During the study, participants will be asked to:

* Follow an early time-restricted eating schedule for one week and their usual eating schedule for another week while keeping to their usual diet and physical activity.
* Attend four visits to the research facility on campus.
* Provide saliva, blood, and urine samples for health marker analysis.
* Complete breathing tests (spirometry and FeNO) to measure lung function.
* Complete short questionnaires about physical activity and quality of life.
* Take part in a short interview about their asthma symptoms and quality of life.
* Keep a brief food diary each week.
* Provide details of any medications they currently take.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18 and 65 years old.
* Control group: individuals without asthma
* Asthma group: Have already been diagnosed with controlled mild asthma.
* Not following any diet regimen.
* Able to read the information pack and give consent in English.

Exclusion Criteria:

* Moderate to severe asthma
* Pregnant
* Smoking
* Systemic corticosteroids.
* History of recent respiratory disease, current chest infection, and collapsed lung.
* History of recent surgery (last 2 months), including thoracic, abdominal, and eye surgery.
* Being diagnosed with cardiovascular diseases, e.g., unstable angina, a heart attack, uncontrolled high blood pressure, stroke, and aneurysm.
* Broken ribs or neck vertebrae.
* Cancer.
* History of autoimmune diseases
* Being diagnosed with an eating disorder.
* Overnight shift work

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Lung Function Parameters, FEV1 in Liters (L) | At baseline and after 1 week in each study arm
  A spirometry test will be conducted to gather information about lung function parameters.
Lung Function Parameters, FVC in Liters (L) | At baseline and after 1 week in each study arm
  A spirometry test will be conducted to gather information about lung function parameters.
Lung Function Parameters, FEV1/ FVC ratio | At baseline and after 1 week in each study arm
  A spirometry test will be conducted to gather information about lung function parameters.
Fractional Exhaled Nitric Oxide (FeNO) in parts per billion (ppb) | At baseline and after 1 week in each study arm
  Fractional exhaled nitric oxide (FeNO) test will be conducted to gather information about airway inflammation.
Blood for health biomarkers | At baseline and after 1 week in each study arm
  Changes in plasma-based health biomarkers will be assessed from acellular plasma extracted from venous blood samples to explore physiological responses to the intervention. Biomarker results will be summarized descriptively.
Urinary Biomarker Profile | At baseline and after 1 week in each study arm
  The urinary metabolomic profile will be assessed to explore changes in metabolites associated with the intervention. Results will be summarized descriptively.
Salivary Metabolomic Profile | At baseline and after 1 week in each study arm
  Salivary metabolomic profile will be assessed to explore changes in metabolites associated with the intervention. Metabolomic features will be summarized descriptively.
body weight in kilograms (Kg) | At baseline and after 1 week in each study arm
  Calibrated electronic scales will be used to measure body weight in kilograms.
Height in meters (m) | At baseline and after 1 week in each study arm
  A stadiometer will be used to measure height in meters.
Demographic Data | At baseline
  Demographic data such as age, sex and ethnicity.

SECONDARY OUTCOMES:
Changes in Quality of Life using Asthma Quality of Life Questionnaire (AQLQ) | At baseline and after 1 week in each study arm
  The Asthma Quality of Life Questionnaire (AQLQ) will be given to assess changes in quality of life in individuals with asthma.
Changes in Quality of Life using PROMIS Global Health v1.2 | At baseline and after 1 week in each study arm
  The PROMIS Global Health v1.2 will be given to assess changes in quality of life for individuals without asthma.
Semi-structured interview for assessing quality of life and acceptability of interventions. | After 1 week of eTRE
  A semi-structured interview will be conducted among participants with mild asthma who are assigned to the eTRE group to assess the challenges they faced and their experiences after the eTRE intervention.

OTHER OUTCOMES:
A Food Diary Record | During the 7-day intervention period (any 3 days)
  A food diary will be given to record and keep track of participants' diet over three consecutive or non-consecutive days, selected by the participants during the 7 days intervention period.
Adherence Monitoring | Before eTRE
  All participants will be given an adherence log to fill out daily as we aim to monitor their adherence. The participant will be reminded every day by email to fill out the log and ensure their adherence to the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Health and Life Science, Leicester, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to institutional policy related to participant confidentiality.